CLINICAL TRIAL: NCT01611064
Title: A Randomised Controlled Trial to Investigate Whether Oxygen Supplementation Can Extend the Time Tolerated or Reduce the Pain Associated With an Upper Limb Tourniquet for Hand Surgery Under Local Anaesthetic
Brief Title: A Study Investigating Ways to Make Local Anaesthetic Hand Surgery Less Painful - Reducing Tourniquet Associated Pain
Acronym: ReTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, Natalia White, BA BMBCh, Senior House Officer in Plastic Surgery, Principle Investigator, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ReTAP Study
Record Dates: First submitted 2012-05-24; First posted 2012-06-04 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hand Injuries/Disease Requiring Surgery to the Hand
Keywords: Hand; Surgery; Tourniquet; Pain; Oxygen
MeSH Terms: conditions — Hand Injuries; Pain | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Active Comparator): Volunteer receives oxygen at a rate of 10litres/minute by mask
  Interventions: Drug: Oxygen
- Air (Placebo Comparator): Volunteer receives normal air at a rate of 10litres/minute by mask
  Interventions: Drug: Medical air

INTERVENTIONS:
Drug: Oxygen — Pure oxygen delivered by simple adult oxygen mask at rate of 10 litres/minute. Commencing 3 minutes prior to tourniquet inflation and administered for a maximum of 45 minutes
  Other Names: O2
  Arms: Oxygen
Drug: Medical air — Pure medical air (21% oxygen content) delivered by simple adult oxygen mask at rate of 10 litres/minute. Commencing 3 minutes prior to tourniquet inflation and administered for a maximum of 45 minutes
  Other Names: Room air; Piped air
  Arms: Air

SUMMARY:
Hand surgery requires a reduced blood flow to the hand during the operation, which is achieved using a tourniquet (tightly inflated circumferential cuff) around the upper arm. However this tourniquet is painful. This study investigates whether breathing oxygen can reduce the pain associated with the tourniquet to both improve patient experience and potentially to allow longer operations to be completed under a local anaesthetic (rather than a general anaesthetic, where the patient is put to sleep, which is more costly, time consuming and risky for the patient).

DETAILED DESCRIPTION:
* This study is a randomised controlled trial of healthy volunteers (for example medical students, nurses and doctors).
* Each volunteer is randomised to receive either oxygen or normal air through a mask whilst wearing an inflated upper arm tourniquet and rating their pain on a scale. The equipment set-up is identical for each volunteer, with the tourniquet inflated to a pressure of 250mmHg in every person.
* Within each arm of the study, volunteers are again randomised to wear the tourniquet on either their dominant or non-dominant arm.
* The study is double-blind (the volunteer and the investigator running the test are unaware of whether oxygen or air is being received) to avoid bias.
* The volunteer can ask for the tourniquet to be removed at any time and will wear the tourniquet for a maximum of 30 minutes.
* The pain ratings and also heart rate and blood pressure are then analysed to identify whether the volunteers receiving oxygen experienced less pain or were able to tolerate the tourniquet for longer than those receiving air.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* More than 18 years of age

Exclusion Criteria:

* Diabetes
* Vascular disease
* Previous operations to arms
* Raynaud's disease
* Analgesia taken in last 24 hours
* Chronic pain
* Hypertension
* Allergy to any substance used in the study
* Unable to give valid consent to participate
* Obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale pain score with time | At 2 minute intervals for a total duration of 45 minutes

SECONDARY OUTCOMES:
Heart rate | Every 6 minutes for a total duration of 45 minutes
Blood pressure | Every 6 minutes for a total duration of 45 minutes
Oxygen saturations | Every 6 minutes for a total duration of 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Natalia White, BA BMBCh, Principal Investigator — Oxford University Hospitals Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] White N, Dobbs TD, Murphy GRF, Khan K, Batt JP, Cogswell LK. Oxygen reduces tourniquet-associated pain: a double-blind, randomized, controlled trial for application in hand surgery. Plast Reconstr Surg. 2015 Apr;135(4):721e-730e. doi: 10.1097/PRS.0000000000001028. PMID 25811584